CLINICAL TRIAL: NCT00094913
Title: Clinical Correlates of Longitudinal PET Changes in Alzheimer's Disease (AD)
Brief Title: PET Changes in Alzheimer's Disease (AD)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Other Study IDs: IA0055; R01AG013616 (NIH)
Record Dates: First submitted 2004-10-28; First posted 2004-10-29 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2007-07

CONDITIONS: Alzheimer Disease
Keywords: Aging; Mild Cognitive Impairment; Alzheimer disease, preclinical; Hippocampal formation; Glucose metabolism
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to identify the earliest predictors of memory and brain deterioration in pre-clinical Alzheimer's disease using positron emission tomography (PET) to monitor brain glucose metabolism.

DETAILED DESCRIPTION:
Previous studies indicate that the brain's glucose metabolism rate potentially may be an early indicator of damage to particular regions of the brain caused by AD, including loss of neurons, synapses, and other changes. Many of these changes are reported among patients with mild cognitive impairment (MCI), a group known to be at increased risk for AD.

The overall goal of this study is to use FDG-PET (2-[(18)F]fluoro-2-deoxy-d-glucose/positron-emission tomography) to determine whether metabolic abnormalities in the hippocampus predict memory and brain deterioration in middle age, and to identify the brain glucose metabolism predictors of future MCI.

Participants in the study will be grouped into 3 main groups of 35 each, including young individuals (20-40 years of age), 41-90 year-old normal, and MCI individuals with or without risk for memory decline. Participants will undergo baseline and 36-month follow-up exams to include comprehensive medical, neurologic, and psychiatric evalutions; lumbar puncture; a resting FDG-PET; an MRI scan; and a neuropsychological battery. A brief medical exam, full neuropsychological battery, and MRI scan will be administered at 18 months. Two subgroups (groups 4 and 5) of 15 each will be created from groups 1 and 2 at 18 months to participate in the evaluation of memory performance under acute hyperglycemia and saline challenges and effects on hippocampal formation and glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with a minimum high school education and between the ages of 50 and 90 will be selected for Groups 1 and 2. For Group 3, normal subjects between the ages of 20 and 49 years of age will be selected. The Groups 1 and 2 will be balanced for age, and all three groups balanced for gender and ApoE genotype.
* Discontinuance of all psychotropic and/or cognitively active medication at least four weeks prior to evaluation.

Exclusion Criteria:

* Past history or MRI evidence of brain damage including significant trauma, stroke, hydrocephalus, lacunar infarcts, seizures, mental retardation or serious neurological disorder.
* Significant history of alcoholism or drug abuse.
* Any history of psychiatric illness (e.g., schizophrenia, mania or depression).
* Any focal signs or significant neuropathology.
* A score of 4 or greater on the Modified Hachinski Ischemia Scale, indicative of cerebrovascular disease.
* A total score of 16 or more on the Hamilton Depression Scale to exclude possible cases of primary depression.
* Evidence of clinically relevant hypertensive, cardiac, pulmonary, vascular, metabolic or hematologic conditions. Specific exclusion will be made for individuals with fasting glucose levels >110 mg/dl.
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Hostility or refusal to cooperate.
* Any prosthetic devices (e.g., pacemaker or surgical clips) that could be affected by the magnetic field employed during MRI imaging.
* Evidence of cognitive or memory impairment reaching early AD levels at the initial evaluation. At baseline, delayed paragraph recall z-scores > 2 below the reference group.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2004-05; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Mony J. de Leon, Ed.D., Principal Investigator — Center for Brain Health, Silberstein Institute
Locations (1):
- Center for Brain Health, Silberstein Institute, New York University, New York, New York, United States

REFERENCES:
- [Background] de Leon MJ, Convit A, Wolf OT, Tarshish CY, DeSanti S, Rusinek H, Tsui W, Kandil E, Scherer AJ, Roche A, Imossi A, Thorn E, Bobinski M, Caraos C, Lesbre P, Schlyer D, Poirier J, Reisberg B, Fowler J. Prediction of cognitive decline in normal elderly subjects with 2-[(18)F]fluoro-2-deoxy-D-glucose/poitron-emission tomography (FDG/PET). Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10966-71. doi: 10.1073/pnas.191044198. Epub 2001 Aug 28. PMID 11526211
- [Background] Bobinski M, de Leon MJ, Convit A, De Santi S, Wegiel J, Tarshish CY, Saint Louis LA, Wisniewski HM. MRI of entorhinal cortex in mild Alzheimer's disease. Lancet. 1999 Jan 2;353(9146):38-40. doi: 10.1016/s0140-6736(05)74869-8. No abstract available. PMID 10023955
- [Background] De Santi S, de Leon MJ, Rusinek H, Convit A, Tarshish CY, Roche A, Tsui WH, Kandil E, Boppana M, Daisley K, Wang GJ, Schlyer D, Fowler J. Hippocampal formation glucose metabolism and volume losses in MCI and AD. Neurobiol Aging. 2001 Jul-Aug;22(4):529-39. doi: 10.1016/s0197-4580(01)00230-5. PMID 11445252